CLINICAL TRIAL: NCT04070300
Title: Physical Activity and Ventricular Arrhythmias
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018/1592
Record Dates: First submitted 2019-08-21; First posted 2019-08-28 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Tachycardia, Ventricular; Defibrillators, Implantable
Keywords: Exercise Training
MeSH Terms: conditions — Tachycardia, Ventricular | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interval training group (Experimental): Aerobic interval training during 12 weeks 3 times a week.
  Interventions: Behavioral: Interval exercise
- Control group (No Intervention): No lifestyle recommendations. Usual daily life.

INTERVENTIONS:
Behavioral: Interval exercise — Aerobic interval training during 12 weeks 3 times a week: 4 x 4 minutes intervals at an intensity of 90-95% of VO2 peak and active breaks of 3 minutes between intervals.
  Other Names: interval training; aerobic exercise training
  Arms: Interval training group

SUMMARY:
The purpose of the study is to determine the effect of aerobic interval training in patients with an implantable cardioverter defibrillator (ICD) on physical fitness, quality of life and the amount of serious ventricular arrhythmic events on short and long term.

DETAILED DESCRIPTION:
In this study, participants will be randomly assigned to either take part in the exercise program or serve as control and live as usual. At baseline study visit, study researchers will review medical records to collect various information, including the reason for needing an ICD, the type and settings of the ICD, medication use and medical history etc. All participants will undergo blood collection, complete a questionnaire to assess quality of life and undergo examination with echocardiography and ECG. The ICD will be programmed accordingly to international guidelines regarding ICD-therapy and optimal monitoring, before each participant complete an exercise treadmill test to determine VO2 peak. They will wear a Holter monitor to record heart activity 48 hours before the test and 24 hours after the test. All participants will then be observed for 2 months before being randomly assigned to either intervention or control. During this observation period, they will wear a fitness activity tracker wristband to evaluate degree of physical activity and a Holter monitor to register number of premature ventricular contractions. Participants taking part in the interval training group will perform aerobic interval training 4 x 4 minutes intervals, 3 times a week for 12 weeks (week 1-12), whereas participants taking part in the control group will carry on with usual daily life with no lifestyle recommendations. All participants will then undergo a new period of observation (week 13-20) and repeat the tests and examinations performed at baseline and during the observation period prior to intervention/control.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ICD and dilated cardiomyopathy or coronary heart disease as cause for implantation
* ICD implanted at St Olavs hospital, Trondheim

In case of difficulties with patient inclusion for the study, the criteria might be broadened to include patients with idiopathic ventricular arrhythmia as cause for implantation.

Exclusion Criteria:

* inability to accomplish the exercise program due to serious comorbidity or to participate in regular training within the next 3 months due to other reasons
* signs of severe cardiac ischemia or persistent ventricular tachycardia during individualized treadmill O2 peak test, which after individual assessment is to be found at risk
* comorbidity where endurance training at more than moderate intensity is discouraged
* severe cardiac valve disease
* planned surgery within the next 3 months
* inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2022-09-02 (Actual)

PRIMARY OUTCOMES:
Change in physical fitness/aerobic capacity | Change from baseline and after ended intervention period (12 weeks)
  Expressed in and measured with maximal oxygen uptake (VO2 peak)
Change in assessment of quality of life | Change from baseline and after intervention period (12 weeks)
  Patient-reported survey of patient health SF-36

SECONDARY OUTCOMES:
Change in burden of ventricular arrhythmias from baseline to week 9-12 | Baseline and the last 4 weeks of intervention period (week 9-12)
  Evaluated by number of ICD discharges (registered on ICD)
Change in burden of ventricular arrhythmias from baseline to week 13-16 | Baseline and the first 4 weeks after intervention period (week 13-16)
  Evaluated by number of ICD discharges (registered on ICD)
Change in burden of ventricular arrhythmias from baseline to week 9-16 | Baseline and the last 4 weeks of intervention period plus 4 first weeks after intervention period (week 9-16)
  Evaluated by number of ICD discharges (registered on ICD)
Change in burden of ventricular arrhythmias from baseline to week 9-12 | Baseline and the last 4 weeks of intervention period (week 9-12)
  Evaluated by number of episodes with antitachycardia pacing (registered on ICD)
Change in burden of ventricular arrhythmias from baseline to week 13-16 | Baseline and the first 4 weeks after intervention period (week 13-16)
  Evaluated by number of episodes with antitachycardia pacing (registered on ICD)
Change in burden of ventricular arrhythmias from baseline to week 9-16 | Baseline and the last 4 weeks of intervention period plus 4 first weeks after intervention period (week 9-16)
  Evaluated by number of episodes with antitachycardia pacing (registered on ICD)
Change in burden of ventricular arrhythmias from baseline to week 9-12 | Baseline and the last 4 weeks of intervention period (week 9-12)
  Evaluated by number of episodes with monitored ventricular tachycardias without ICD-therapy (registered on ICD)
Change in burden of ventricular arrhythmias from baseline to week 13-16 | Baseline and the first 4 weeks after intervention period (week 13-16)
  Evaluated by number of episodes with monitored ventricular tachycardias without ICD-therapy (registered on ICD)
Change in burden of ventricular arrhythmias from baseline to week 9-16 | Baseline and the last 4 weeks of intervention period plus 4 first weeks after intervention period (week 9-16)
  Evaluated by number of episodes with monitored ventricular tachycardias without ICD-therapy (registered on ICD)
Change in burden of ventricular arrhythmias from baseline to week 9-12 | Baseline and the last 4 weeks of intervention period (week 9-12)
  Evaluated by number of premature ventricular contractions (registered on a 72 hours Holter monitoring)
Change in burden of ventricular arrhythmias from baseline to week 13-16 | Baseline and the first 4 weeks after intervention period (week 13-16)
  Evaluated by number of premature ventricular contractions (registered on a 72 hours Holter monitoring)
Change in burden of ventricular arrhythmias from baseline to week 9-16 | Baseline and the last 4 weeks of intervention period plus 4 first weeks after intervention period (week 9-16)
  Evaluated by number of premature ventricular contractions (registered on a 72 hours Holter monitoring)
Cardiac function | Baseline and after ended intervention period (12 weeks)
  Evaluated by changes in left ventricular dimensions and systolic/diastolic function assessed by echocardiography and blood values (NT-proBNP and troponin T)
Change in degree of physical activity | Baseline and after ended intervention period (12 weeks)
  Assessed by number of steps daily registered with fitness activity tracker wristband (worn for 1 week)
Changes in adiposity | Baseline and after ended intervention period (12 weeks)
  Evaluated by changes in waist circumference (cm) and BMI (kg/m^2) as measures of adiposity
Changes in cholesterol value | Baseline and after ended intervention period (12 weeks)
  Evaluated by changes in total cholesterol, HDL-cholesterol, LDL-cholesterol (all in mmol/L) as a measure of cardiac risk
Changes in triglycerides value | Baseline and after ended intervention period (12 weeks)
  Evaluated by changes in triglycerides ( in mmol/L) as a measure of cardiac risk
Changes in heart rate variability | Baseline and after ended intervention period (12 weeks)
  Evaluated by measuring changes in SDNN, SDANN 5, ASDNN 5 and RMSSD registered on a 72 hours Holter monitoring
Changes in number of premature ventricular contractions during a single bout of high intensity exercise (VO2 peak test) | Baseline and after ended intervention period (12 weeks)
  Measured by changes in the number of premature ventricular contractions during VO2 peak testing
Changes in signal-averaged ECG (SA-ECG) | Baseline and after ended intervention period (12 weeks)
  Measured by quantifying late potentials after depolarization of the ventricles

CONTACTS AND LOCATIONS:
Overall Officials: Rune Wiseth, MD, Prof, Study Director — St. Olavs Hospital
Locations (1):
- St Olavs Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data for all primary and secondary outcome measures will be made available after deidentiﬁcation and publication
Time Frame: After publication
Access Criteria: Not yet decided